CLINICAL TRIAL: NCT07183709
Title: Phase 1 Dose Ranging Study to Assess the Safety, Reactogenicity, and Immunogenicity of PepGNP-COVID19, a Synthetic Nanoparticle-based, T Cell Priming Peptide Vaccine Against SARS-CoV-2 As a Booster Dose
Brief Title: Safety and Immunogenicity Trial of PepGNP-COVID19 Vaccine in Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 25-1105
Record Dates: First submitted 2025-09-18; First posted 2025-09-19 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01-09

CONDITIONS: COVID-19
Keywords: booster dose; Covid-19; Dose Ranging; Immunogenicity; PepGNP-COVID19; Phase 1; Reactogenicity; Safety; SARS-CoV-2; Vaccine
MeSH Terms: conditions — COVID-19 | interventions — Injections

STUDY DESIGN:
Who Masked: Participant
Masking Description: This study will be single blinded. Participants will be blinded to the dose of the study product that they receive, to reduce potential bias in reporting reactogenicity and adverse events (AEs). Since the three doses of the PepGNPCovid19 vaccine are of the same volume and appearance, no masking of the Nanopass MicronJet (TM) 600 delivery device is needed. Participants will be unblinded and informed of the dose of the study product they received at the final study visit, following institutional policies. Study personnel performing immunogenicity assays will be blinded.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Experimental): 0.05ml of 0.83nmol PepGNP-COVID19 administered intradermally on Day 1 in Healthy Adult participants, 18 to 64 years of age; (8 of 20 participants aged > / = 50 years) N= 20
  Interventions: Biological: PepGNP-COVID19; Other: Sterile Water for Injection
- Cohort 2 (Experimental): 0.05ml of 2.5nmol PepGNP-COVID19 administered intradermally on Day 1 in Healthy Adult participants, 18 to 64 years of age; (8 of 20 participants aged > / = 50 years) N= 20
  Interventions: Biological: PepGNP-COVID19; Other: Sterile Water for Injection
- Cohort 3 (Experimental): 0.05ml of 7.5 nmol PepGNP-COVID19 administered intradermally on Day 1 in Healthy Adult participants, 18 to 64 years of age; (8 of 20 participants aged > / = 50 years) N= 20
  Interventions: Biological: PepGNP-COVID19; Other: Sterile Water for Injection

INTERVENTIONS:
Biological: PepGNP-COVID19 — A synthetic T cell priming setpoint-modifying SARS-CoV-2 vaccine composed of ultrasmall carbohydrate-coated gold nanoparticles carrying covalently bound MHC class I-binding SARS-CoV-2 peptides.
Other: Sterile Water for Injection — A sterile, nonpyrogenic preparation of water for injection which contains no bacteriostat, antimicrobial agent or added buffer and is supplied only in single-dose containers to dilute or dissolve drugs for injection

SUMMARY:
This Phase 1 clinical trial will evaluate the safety, reactogenicity, and immunogenicity of PepGNP-COVID19, a synthetic nanoparticle-based, T cell-priming peptide vaccine against SARS-CoV-2, when administered as a booster dose in healthy adults. PepGNP-COVID19 is designed to induce broad and durable T cell-mediated immune responses by delivering conserved SARS-CoV-2 peptides covalently bound to carbohydrate-coated gold nanoparticles, with the goal of enhancing tissue-resident cytotoxic T lymphocytes in the respiratory tract and reducing the need for frequent antigen updates. This randomized, participant-blinded, dose-ranging, multi-site trial will enroll 60 healthy adults aged 18-64 years, with a target of 8 of 20 participants in each cohort being > / = 50 years of age. Participants will receive a single intradermal injection of PepGNP-COVID19 at one of three dosage levels (0.83 nmol, 2.5 nmol, or 7.5 nmol in a volume of 0.05 mL).

The primary objective is to evaluate the safety, reactogenicity, and tolerability of a single intradermal dose of PepGNP-COVID19 at three dosage levels in previously vaccinated healthy adults.

DETAILED DESCRIPTION:
This Phase 1 clinical trial will evaluate the safety, reactogenicity, and immunogenicity of PepGNP-COVID19, a synthetic nanoparticle-based, T cell-priming peptide vaccine against severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), when administered as a booster dose in healthy adults. PepGNP-COVID19 is designed to induce broad and durable T cell-mediated immune responses by delivering conserved SARS-CoV-2 peptides covalently bound to carbohydrate-coated gold nanoparticles. The goal is to enhance tissue-resident cytotoxic T lymphocytes in the respiratory tract and reduce the need for frequent antigen updates. This is a randomized, participant-blinded, dose-ranging, multi-site trial in healthy adults 18-64 years of age, with a target of 8 of 20 participants in each cohort being > / = 50 years of age. A total of 60 participants will be enrolled, with 20 participants assigned to each cohort. Participants will receive a single intradermal injection (ID) of PepGNP-COVID19 at one of three dose levels: 0.83 nmol, 2.5 nmol, or 7.5 nmol in a volume of 0.05 mL.

The primary objective is to evaluate the safety, reactogenicity, and tolerability of a single intradermal dose of PepGNP-COVID19 at three dosage levels in previously vaccinated healthy adults, as assessed by: a) Solicited local and systemic adverse events (AEs) through 7 days after vaccination; b) Unsolicited AEs through 28 days after vaccination; c) Abnormal clinical safety laboratory AEs through 14 days after vaccination; d) Serious adverse events (SAEs), medically attended adverse events (MAAEs), new-onset chronic medical conditions (NOCMCs), adverse events of special interest (AESIs), and potentially immune-mediated diseases (pIMDs) through 6 months after vaccination; e) Vaccine tolerability assessment on Day 29. The secondary objectives are to assess systemic T cell-mediated immune responses and to evaluate systemic anti-Spike humoral immune responses following a single ID of PepGNP-COVID19.

ELIGIBILITY:
Inclusion Criteria:

1. Provides written informed consent prior to initiation of any study procedures.
2. Able to understand and agrees to comply with planned study procedures and be available for all study visits.
3. Non-pregnant adults, 18 through 64 years of age, inclusive at time of study product administration.
4. Participants of childbearing potential* must agree to use or have practiced true abstinence** or use at least one acceptable primary form of contraception*** *These criteria apply to females who are in a heterosexual relationship who are of childbearing potential. Not of childbearing potential include post-menopausal females (defined as having a history of amenorrhea for at least one year) or a documented status as being surgically sterile (hysterectomy, bilateral oophorectomy, or tubal ligation/salpingectomy).

   **True abstinence is 100% of the time, no sexual intercourse (penis enters the vagina). Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods.

   ***Acceptable forms of primary contraception include a monogamous relationship with a vasectomized partner who has been vasectomized for 180 days or more before the participant's study product administration, intrauterine devices, birth control pills, and injectable/implantable/insertable/transdermal hormonal birth control products. Must have used at least one acceptable primary form of contraception for at least 30 days before study product administration and agree to continue at least one acceptable primary form of contraception through 60 days after study product administration.
5. Participants of childbearing potential must have a negative urine pregnancy test at screening and within 24 hours prior to study product administration.
6. In general self-reported, good health.****

   ****As determined by medical history and physical examination, including vital signs, to evaluate acute or ongoing chronic medical diagnoses/conditions that have been present for at least 90 days, which would affect the assessment of the safety of participants. Chronic medical diagnoses/conditions should be stable for the last 30 days (i.e., no hospitalizations, ER, or urgent care for the condition). This includes no change in chronic prescription medication, dose, or frequency due to deterioration of the chronic medical diagnosis/condition 30 days before the study product administration. Any prescription change due to a change of health care provider, insurance company, etc., or done for financial reasons and in the same class of medication will not be considered a deviation of this inclusion criterion. Participants may be on chronic or as-needed (prn) medications if, in the opinion of the participating site PI or appropriate sub-investigator, they pose no additional risk to participant safety or assessment of reactogenicity and immunogenicity.
7. Receipt of a complete primary authorized or approved COVID-19 vaccine series and at least one booster***** with last vaccination at least 16 weeks prior to study product administration.

   *****Primary series and/or booster may have been received as part of participation in a clinical trial (see MOP for further details).
8. Clinical screening laboratory evaluations are within normal reference ranges or grade 1 with no clinical significance (NCS) per investigator discretion.
9. Must agree to have samples stored for secondary research.

Exclusion Criteria:

1. Positive SARS-CoV-2 Polymerase Chain Reaction [PCR] at screening.
2. Abnormal vital signs at screening (Grade 1 or higher) *:

   *Grade 1 or higher is equivalent to: Systolic blood pressure (SBP) > / =141 mmHg or < / = 89 mmHg Diastolic blood pressure (DBP) > / =91 mmHg Heart rate (HR) is > / =101 beats per minute or < / = 54 beats per minute Oral temperature > / =38.0°C (100.4°F)
3. History of SARS-CoV-2 infection or receipt of any COVID-19 vaccine < 16 weeks prior to study product administration.
4. Pregnant or breastfeeding.
5. Blood or plasma donation within 4 weeks prior to planned study product administration.
6. Receipt of antibody or blood-derived products within 90 days prior to planned study product administration.
7. Any self-reported or documented significant medical or psychiatric diseases** or any other condition that, in the opinion of the site PI or appropriate sub-investigator, precludes study participation.

   **Significant medical or psychiatric conditions include but are not limited to significant kidney disease, liver disease, history of hematologic malignancy, ongoing other malignancy or recent diagnosis of malignancy in the last five years excluding treated basal cell and squamous cell carcinoma of the skin, and cervical carcinoma in situ, which are allowed.
8. History of any significant neurological or neurodevelopmental conditions.***

   ***Including history of Bell's palsy, history of four or more migraine headaches in the past 12 months that interfered with normal daily activity or any migraine headache in the past 5 years that required emergency or inpatient medical care, epilepsy, seizures in the last 5 years, encephalopathy, focal neurologic deficits, Guillain-Barré syndrome, encephalomyelitis, transverse myelitis, stroke or transient ischemic attack, multiple sclerosis, Parkinson's disease, amyotrophic lateral sclerosis, Creutzfeldt-Jakob disease, or Alzheimer's disease.
9. History of significant respiratory disease requiring daily medications currently, history of asthma in the past 5 years, or any treatment of respiratory disease exacerbations in the last 5 years.
10. History of cardiovascular disease (e.g., congestive heart failure, cardiomyopathy, ischemic heart disease), including any history of myocarditis or pericarditis, or uncontrolled cardiac arrhythmia.
11. Any autoimmune disease, including hypothyroidism, without a defined non-autoimmune cause.
12. Has an acute illness, as determined by the site PI or appropriate sub-investigator within 72 hours prior to study product administration.****

    ****An acute illness that is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the participating site PI or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.
13. Has a positive test result for hepatitis B surface antigen, hepatitis C virus RNA (by reflex testing), or human immunodeficiency virus (HIV) antigen/antibody test at screening.
14. Has any confirmed or suspected immunosuppressive or immunodeficient state such as asplenia, recurrent severe infections, or chronic***** immunosuppressant medication within the past 6 months or is planning to receive one during the study.******

    *****Chronic means more than 14 continuous days.

    ******Topical, ophthalmic, inhaled, and intraarticular corticosteroids are acceptable, but receipt of =20 mg/day of prednisone or equivalent for =14 consecutive days in the 4 weeks prior to signing ICF is exclusionary. See exclusion 19 for intranasal steroids.
15. Has received any investigational study product within 60 days, or 5 half-lives, whichever is longer, before study product administration or is planning to receive one during the study.
16. Has a history of hypersensitivity or severe allergic reaction******* to any previous licensed or unlicensed vaccine or the candidate vaccine components (e.g., gold).********

    *******(e.g., anaphylaxis, generalized urticaria, angioedema, other significant reaction)

    ********See IB for vaccine formulation.
17. Received or plans to receive licensed inactivated/subunit vaccine within 14 days of study product administration or live vaccine within 28 days of study product administration.
18. Plan to receive a COVID-19 booster vaccine within the 180 days following study product administration.
19. Regular use of intranasal medications, including steroids.*********

    *********Participant must have had no intranasal medication use for 30 days prior to study product administration and plans not to use intranasal medications for 30 days after study product administration for medications other than steroids, and for 3 months after study product administration for intranasal steroids (including over-the-counter [OTC] medications such as Flonase).
20. Use of intranasal illicit drugs in the 5 years prior to study product administration or plans to use during the study.
21. Current smoker (including cigarettes, marijuana, and vaping) or smoking within the prior 3 months.
22. History of keloid formation.
23. Current or past scars, tattoos, or other disruptions of skin integrity at the intended site of study product administration that would preclude adequate assessment of injection site reactogenicity.
24. History of alcohol or illicit drug abuse within 6 months of enrollment that, in the opinion of the site PI or appropriate sub-investigator, precludes study participation.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-10-20 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants experiencing Abnormal Clinical Safety Laboratory Adverse Events | Day 1 through Day 14
Proportion of participants experiencing Adverse Events of Special Interest (AESI) | Day 1 through Day 180
Proportion of participants experiencing Medically Attended Adverse Events (MAAEs) | Day 1 through Day 180
Proportion of participants experiencing New Onset Chronic Medical Conditions (NOCMCs) | Day 1 through Day 180
Proportion of participants experiencing potentially immune-mediated diseases (pIMDs) | Day 1 through Day 180
Proportion of participants experiencing Serious Adverse Events (SAEs) | Day 1 through Day 180
Proportion of participants experiencing Solicited Local Adverse Events (AEs) | Day 1 through Day 7
Proportion of participants experiencing Solicited Systemic Adverse Events (AEs) | Day 1 through Day 7
Proportion of participants experiencing Unsolicited Adverse Events (AEs) | Day 1 through Day 28
Vaccine tolerability assessment score | Day 29
  Based on responses to Global Tolerability Assessment questionnaire

SECONDARY OUTCOMES:
Level of serum binding antibodies to SARS-CoV-2 Spike variants | Day 1 through Day 181
Percentage of CD8+ T cells specific to vaccine dextramers | Day 1 through Day 181

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Alabama at Birmingham School of Medicine - Infectious Disease, Birmingham, Alabama
  - George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - Cincinnati Children's Hospital Medical Center Vaccine Research Center, Cincinnati, Ohio